CLINICAL TRIAL: NCT04585074
Title: Prospective Cohort Study of Mastectomy With Reconstruction Including Robot Endoscopic Breast Surgery
Brief Title: Prospective Study of MAstectomy With Reconstruction Including Robot Endoscopic Surgery
Acronym: MARRES
Status: Active, not recruiting | Type: Observational
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyung Seok Park, MD, PhD, Professor, Severance Hospital
Other Study IDs: 4-2020-0165
Record Dates: First submitted 2020-09-18; First posted 2020-10-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Breast Neoplasms; Germline BRCA1 Gene Mutation; Germline BRCA2 Gene Mutation; Benign Breast Disease; Germline Mutation Abnormality
Keywords: minimal invasive procedure; robot assisted nipple sparing mastectomy; breast immediate reconstruction; breast neoplasms
MeSH Terms: conditions — Breast Neoplasms; Cystic Fibrosis | interventions — Robotics; Mastectomy, Simple; Mastectomy; Mastectomy, Subcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Robotic or endoscopic nipple sparing mastectomy — Cases or Patients who underwent robotic nipple-sparing mastectomy and immediate reconstruction are enrolled in this arm. Robotic nipple-sparing mastectomy should be performed using robotic surgical systems. Robotic surgical systems include da Vinci S,Si, X, Xi, and SP systems. Axillary or lateral incisions are used for this procedure. Immediate reconstruction includes tissue expander insertion, direct-to-implant, latissimus dorsi flap, transverse abdominis rectus muscle flap, or deep inferior epigastric perforators flap. Cases with robotic mastectomy without immediate reconstruction are excluded.
  Other Names: Robot-assisted nipple sparing mastectomy; Robot mastectomy; Robotic mastectomy; Hybrid robotic nipple sparing mastectomy; Robot-assisted nipple areolar complex and skin sparing mastectomy; Endoscopic nipple sparing mastectomy
Procedure: Conventional mastectomy (including nipple sparing mastectomy, skin sparing mastectomy) — Cases or Patients who underwent conventional mastectomy and immediate reconstruction are enrolled in this arm. Conventional mastectomy should not be performed using robotic or endoscopic surgical systems. Any incisions can be performed for this procedure. Conventional mastectomy includes also Nipple-sparing mastectomy and Skin sparing mastectomy. Immediate reconstruction includes tissue expander insertion, direct-to-implant, latissimus dorsi flap, transverse abdominis rectus muscle flap, or deep inferior epigastric perforators flap. Cases without immediate reconstruction are excluded.
  Other Names: Total mastectomy; Mastectomy; Nipple-sparing mastectomy; Skin sparing mastectomy

SUMMARY:
Robotic mastectomy and immediate reconstruction have been introduced in 2015. However, since robotic mastectomy is the latest surgical technique, there is a lack of studies prospectively comparing conventional mastectomy and immediate reconstruction with robotic mastectomy. For this reason, this study is designed to establish a single institution cohort study that prospectively collects patients undergoing mastectomy and reconstruction. This study was initially designed as a single institution study, however, currently, the study was extended to the multicenter study including 18 institutions over the country. Using the established prospective cohort data, a comparative study of robotic mastectomy with conventional mastectomy and reconstruction, and cost-effectiveness and satisfaction of robotic endoscopic surgery, and cost-effectiveness and satisfaction of reconstructive surgery are to be analyzed.

DETAILED DESCRIPTION:
This study is a multi-institution cohort study that prospectively collects patients undergoing mastectomy and reconstruction.

Patients' inclusion criteria is as below; adult women between the ages of 19 and 80, with breast cancer or high risk of breast cancer (patients with a BRCA1/2 mutation, TP53 mutation, PALB2 mutation, etc) scheduled for therapeutic or prophylactic mastectomy, and want immediate reconstruction.

Patients planned for breast-conserving surgery or who do not want immediate reconstruction will be excluded. Patients who planned for surgery on both sides in the different methods (e.g. right for RNSM and left for conventional open NSM) are also excluded. Meanwhile, cases with ipsilateral NSM and contralateral partial mastectomy or excision are included.

The goal number of enrolled patients is 2000.

Collecting data includes patients' clinicopathological factors including height, weight, etc. And also collecting surgical results, oncological results, cost-effectiveness, and satisfactions of patients to secure high-level data.

The satisfaction of patients using the Breast Q survey, basic characteristics like height, weight, etc, and patients' photos will be collected preoperatively.

Also, patients' data will be collected within 6 months after surgery including clinical-pathological factors, surgery results (drainage amount, removal date, complications), postoperative recovery evaluation, complications and adverse reactions, cost, etc.

Between 6 months and 1 year(Patients who have undergone skin sparing mastectomy can do within up to 3 years) after surgery, the results of surgery, recurrence, satisfaction survey, and postoperative photos will be collected.

Every 12 months thereafter, whether adjuvant therapy (chemotherapy, radiation therapy, targeted therapy, endocrine therapy) was implemented, surgical results, and recurrence will be investigated and collected until the end of the study period.

An interim analysis will be done after completing the recruitment of subjects by the 4th year after the start of the study and collecting data. Complete the follow-up observation and data collection of the subjects recruited in the 5-9 years and the final analysis will be conducted.

Categorial variables will be examined by the chi-square test or Fisher's exact test.

Continuous variables will be examined by t-test or ANOVA, and M-W test or K-W test if needed.

Survival analysis will be examined by Kaplan-Meier plot and log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* Female patient between the ages of 19 and 80
* Patients with breast cancer or high risk of breast cancer ( BRCA1/2 mutation, TP53 mutation, PALB2, etc.)
* Patients scheduled for therapeutic or prophylactic mastectomy (including conventional mastectomy, skin sparing mastectomy, areolar conserving mastectomy)
* Patients who want immediate reconstruction during mastectomy
* Those agreed in writing consent to participate study

Exclusion Criteria:

* Patients scheduled for breast conserving mastectomy
* Patients who do not want immediate reconstruction during mastectomy
* Patients who planned for surgery on both sides in the different methods

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who underwent nipple-sparing mastectomy between 2020 and 2024 at Severance Hospital, Seoul, Korea
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2030-04-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication rates in 30 days | Postoperative 30 days
  Postoperative complication rates are calculated as total number of postoperative complication cases per total operation cases.
Clavien-Dindo grade of postoperative complications | Postoperative 180 days
  Clavien-Dindo grade of postoperative complications is evaluated. The highest grade of postoperative complications are used for the analysis.

SECONDARY OUTCOMES:
Recurrence free survival (RFS) | Postoperative 5 years
  Events of RFS includes locoregional recurrence, distant recurrence, and death. Contralateral breast cancer and second primary malignancy are considered to be censored data.
Cancer incidence rate | Postoperative 5 years
  cancer incidence rate for those underwent prophylactic mastectomy
Patient's satisfaction (about reconstruction expectations) | within preoperative 4 weeks to operation and within postoperative 6 month to 12 month.(Patients who have undergone skin sparing mastectomy can do within up to 3 years)
  Reconstruction Expectations of Preoperative Short Form. In all scales, higher scores reflect a better outcome.
Patient's satisfaction (about reconstruction results) | within preoperative 4 weeks to operation and within postoperative 6 month to 12 month.(Patients who have undergone skin sparing mastectomy can do within up to 3 years)
  1. Mastectomy Module Pre-and Postoperative Scales Satisfaction with Breasts as assessed by BREAST-Q version 2.0. Higher scores reflect a better outcome.
  2. Reconstruction Module Pre-and Postoperative Scales Satisfaction with abdomen as assessed by BREAST-Q version 2.0 (This scale should only be completed by the patient who has had reconstruction using a transverse rectus abdominis myocutaneous flap(TRAM flap) or deep inferior epigastric perforators flap(DIEP flap). Otherwise, skip it.) Satisfaction with Back as assessed by BREAST-Q version 2.0 (This scale should only be completed by the patient who has had reconstruction using a latissimus dorsi flap. Otherwise, skip it.) Satisfaction with Implants as assessed by BREAST-Q version 2.0 (This scale should only be completed by the patient who has had reconstruction using implants. Otherwise, skip it.) In all scales, higher scores reflect a better outcome.
Surgeon's satisfaction | Postoperative 6 month to 12 month(Patients who have undergone skin sparing mastectomy can do within up to 3 years
  Satisfaction of Surgery assessed by (Plastic)Surgeon(s) Items(1), Response Options(Overall symmetry, postoperative scar, nipple areolar complex symmetry, etc), Range(0-10) The higher scores are, the better an outcome is.
Cost-effectiveness | Postoperative 6 month to 1 year(Patients who have undergone skin sparing mastectomy can do within up to 3 years
  Cost-effectiveness evaluation according to the surgical method, by conducting a questionnaire survey on the subject 6 months to 1 year(Patients who have undergone skin sparing mastectomy up to 3 years) after the last surgery. Evaluation follows the EuroQol five-dimension scale(EQ5D, EQ5D-5L) Korean version questionnaire. In all scales, higher scores reflect a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Seok Park, MD, PhD, Principal Investigator — Severance Hospital
Locations (18):
- South Korea (18):
  - Kosin University Gospel Hospital, Busan, Busan
  - Chungnam National University Sejong Hospital, Sejong, Chungcheongnam-do
  - Kyungpook National University Chilgok Hospital, Daegu, Daegu
  - Wonju Severance Christian hospital, Wŏnju, Gangwon-do
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Yongin Severance Hospital, Yongin-si, Gyeonggi-do
  - Samsung Changwon Medical Center, Changwon, Gyeongsangnam-do
  - The Catholic University of Korea, Incheon ST. Mary's Hospital, Incheon, Incheon
  - Korea University Anam Hospital, Seoul, Seoul
  - Seoul National University Hospital, Seoul, Seoul
  - Soonchunhyang University Hospital, Seoul, Seoul
  - Gangnam Severance Hospital, Seoul, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, Seoul
  - Korea University Guro Hospital, Seoul, Seoul
  - Yonsei University College of Medicine, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul

REFERENCES:
- [Background] Banfield S. A management systems analysis. Caring. 1987 Jul;6(7):45-50. No abstract available. PMID 10283322
- [Derived] Ryu JM, Lee J, Lee J, Ko B, Kim JH, Shin H, Park HS; Korea Robot-endoscopy Minimal Access Breast Surgery Study Group (KoREa-BSG). Mastectomy with Reconstruction Including Robotic Endoscopic Surgery (MARRES): a prospective cohort study of the Korea Robot-Endoscopy Minimal Access Breast Surgery Study Group (KoREa-BSG) and Korean Breast Cancer Study Group (KBCSG). BMC Cancer. 2023 Jun 21;23(1):571. doi: 10.1186/s12885-023-10978-0. PMID 37344780